CLINICAL TRIAL: NCT07387432
Title: Role of Exercise in Functional Capacity of Smokers and Subsequent Development of Chronic Obstructive Pulmonary Disease
Brief Title: Role of Exercise in PRISm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 24-461
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Preserved Ratio Impaired Spirometry (PRISM)
Keywords: Preserved ratio impaired spirometry; PRISm; exercise with telehealth; walking exercise; smoking cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise with telehealth group (Experimental): Participants will attend telehealth physiotherapy class for exercise. Smoking cessation advice will be given
  Interventions: Behavioral: Exercise with telehealth group
- Exercise group (Active Comparator): Participants will exercise with walking. Smoking cessation advice will be given
  Interventions: Behavioral: Exercise group
- No exercise group (Active Comparator): No exercise instruction will be given. Participants are encouraged to exercise. Smoking cessation advice will be given
  Interventions: Behavioral: No exercise group

INTERVENTIONS:
Behavioral: Exercise with telehealth group — Participants will attend telehealth physiotherapy class for exercise. Smoking cessation advice will be given.
  Arms: Exercise with telehealth group
Behavioral: Exercise group — Participants will exercise with walking. Smoking cessation advice will be given
  Arms: Exercise group
Behavioral: No exercise group — No exercise instruction will be given. Participants are encouraged to exercise. Smoking cessation advice will be given
  Arms: No exercise group

SUMMARY:
Preserved Ratio Impaired Spirometry (PRISm) describes individual with spirometry findings of forced expiratory volume (FEV1) and forced vital capacity (FVC) ratio greater than 0.7 but with the FEV1 less than 80% predicted.

While the spirometry findings of individuals with PRISm can be transited into obstructive pattern, remains at PRISm or become normal spirometry, limited evidence is on the role of exercise in the course of PRISm. This study aims to investigate the role of exercise, namely exercise with telehealth and walking exercise, together with smoking cessation advice, would alter the clinical course of PRISm.

DETAILED DESCRIPTION:
The is an open-labelled prospective randomised control trial on individuals with spirometry findings of PRISm. Individuals who are smoker/ ex-smoker will be screened by spirometry. Eligible individuals who fulfill the inclusion and exclusion criteria will be recruited and randomised into exercise with telehealth group, exercise group and no exercise group into 1:1:1 ratio.

The intervention period is 26 weeks and the follow up period is 52 weeks. In the intervention period, individuals will be instructed to exercise accordingly. In exercise with telehealth group, exercise with telehealth will be performed 2 times per week for 1 hour. In exercise group, individuals will be instructed to have exercise with each week's goal was the lowest of three numbers: (1) the average of the most recent 7 days of step counts + 600 steps, (2) the previous goal + 600 steps, or (3) 10,000 steps per day. In no exercise group, no exercise instruction will be given.

Smoking cessation advice and clincial assessment including hospitalisation due to any respiratory or cardiovascular causes, modified Medical Research Council Dyspnea Scale, St George's Respiratory Questionnaire will be assessed in baseline, week 4, 8, 12, 26, 52. Spirometry by Spirodoc and 6 minute walk test will be assessed at baseline, week 12, 26 and 52.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* Smoker/ ex-smoker
* Spirometry shows PRISm, with FEV1/FVC >= 0.7 and FEV1 <80% predicted
* Ambulatory to walk
* Able to give informed consent

Exclusion Criteria:

* Age below 18
* Non-smoker
* Spirometry does not show PRISm/ unable to perform spirometry
* Requires assistance for walking
* Umable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in 6 minute walk test distance | 1 year
  The 6 minute walk test distance will be measured in the start of the study, at 3 months, 6 months and 12 months. The difference will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: King Pui Florence Chan, MD, Principal Investigator — he University of Hong Kong, Queen Mary Hospital
Locations (1):
- The University of Hong Kong, Queen Mary Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No
According to the current ethics approval protocol, the IPD will be stored anonymously and destroyed 3 years after completion of study.

REFERENCES:
- [Result] Hansen H, Bieler T, Beyer N, Kallemose T, Wilcke JT, Ostergaard LM, Frost Andeassen H, Martinez G, Lavesen M, Frolich A, Godtfredsen NS. Supervised pulmonary tele-rehabilitation versus pulmonary rehabilitation in severe COPD: a randomised multicentre trial. Thorax. 2020 May;75(5):413-421. doi: 10.1136/thoraxjnl-2019-214246. Epub 2020 Mar 30. PMID 32229541
- [Result] Wan ES, Balte P, Schwartz JE, Bhatt SP, Cassano PA, Couper D, Daviglus ML, Dransfield MT, Gharib SA, Jacobs DR Jr, Kalhan R, London SJ, Navas-Acien A, O'Connor GT, Sanders JL, Smith BM, White W, Yende S, Oelsner EC. Association Between Preserved Ratio Impaired Spirometry and Clinical Outcomes in US Adults. JAMA. 2021 Dec 14;326(22):2287-2298. doi: 10.1001/jama.2021.20939. PMID 34905031
- [Result] Perez-Padilla R, Montes de Oca M, Thirion-Romero I, Wehrmeister FC, Lopez MV, Valdivia G, Jardim JR, Muino A, B Menezes AM; PLATINO Group. Trajectories of Spirometric Patterns, Obstructive and PRISm, in a Population-Based Cohort in Latin America. Int J Chron Obstruct Pulmon Dis. 2023 Jun 21;18:1277-1285. doi: 10.2147/COPD.S406208. eCollection 2023. PMID 37366430
- [Result] Holland AE, Cox NS, Houchen-Wolloff L, Rochester CL, Garvey C, ZuWallack R, Nici L, Limberg T, Lareau SC, Yawn BP, Galwicki M, Troosters T, Steiner M, Casaburi R, Clini E, Goldstein RS, Singh SJ. Defining Modern Pulmonary Rehabilitation. An Official American Thoracic Society Workshop Report. Ann Am Thorac Soc. 2021 May;18(5):e12-e29. doi: 10.1513/AnnalsATS.202102-146ST. PMID 33929307
- See also: Related Info — https://goldcopd.org/